CLINICAL TRIAL: NCT06661928
Title: Conservative Surgery with Modified Widman Flap Vs Conservative Surgery with Papilla Preservation Technique for the Treatment of Residual Pockets: a 5-year Randomized Clinical Trial
Brief Title: Conservative Surgery with Modified Widman Flap Vs Papilla Preservation Technique for the Treatment of Residual Pockets
Acronym: MWF vs PPT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Mario Aimetti, Associate Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TurinPerioSurgery02
Record Dates: First submitted 2024-10-22; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Papilla preservation flap (Experimental): Access flap for open flap debridement using intrasulcular incisions and papilla preservation approaches to preserve the entire interdental tissues
  Interventions: Procedure: Papilla preservation flap
- Conventional surgery (Active Comparator): Access flap for open flap debridement using a conventional modified Widman flap procedure
  Interventions: Procedure: Widman flap procedure

INTERVENTIONS:
Procedure: Papilla preservation flap — Surgical access will be obtained using modified papilla preservation techniques and when interproximal space is narrow (less than 3mm in width) incision will be made using the simplified papilla preservation flap. Both flaps buccal and lingual/palatal will be elevated in any case to allow root surface cleaning and defects debridement under direct vision. Minimally invasive flap elevation preventing to damage inter proximal tissues with the preservation of the papilla. Defects debridement with mini-curettes. Root surface debridement with ultrasonic debridement with periotip and mini-curettes. Flaps will be positioned at the pre-surgical level without any tension. Monofilament non-resorbable 5-0 e-PTFE suturing material will be used.
  Suturing will be performed with external vertical mattress sutures to achieve primary intention closure.
  Arms: Papilla preservation flap
Procedure: Widman flap procedure — Surgical access will be obtained using the modified Widman flap technique. Intrasulcular incision will be done on both buccal and lingual/palatal sides without attempting to preserve the interdental tissues and interdental tissues will be removed. Both flaps buccal and lingual/palatal will be elevated at full thickness in any case to allow root surface cleaning and defects debridement under direct vision, a vertical releasing incision could be made when needed.
  Defects debridement with mini-curettes. Root surface debridement with ultrasonic debridement with periotip and mini-curettes. Flaps will be positioned at the level of the alveolar crest without tension. Monofilament nonresorbable 5 - 0 e/PTFE suturing material will be used. Suturing will be performed with single interrupted sutures.
  Arms: Conventional surgery

SUMMARY:
The primary aim of the study is to evaluate the efficacy of conservative surgery with or without papilla preservation technique in the treatment of deep residual pockets ≥ 6 mm in stage III-IV periodontitis patients after cause related therapy (step II) in terms of endpoints of therapy and other secondary outcomes at different time intervals (1, 3 and 5 years). Moreover, the study aims to evaluate the stability of the results obtained for the different surgical approaches over a 5 years follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage III/IV periodontitis.
* Completed steps I-II periodontal therapy at least 6 weeks before.
* Full mouth plaque score of less than 15% at re-evaluation.
* Full mouth bleeding score of less than 15% at re-evaluation.
* Sextant with residual probing pocket depth (PPD) ≥ 6 mm at ≥ 2 natural teeth (third molars excluded).
* Signed informed consent.

Exclusion Criteria:

* Compromised general health which contraindicates the study procedures (ASA III-VI patients).
* Systemic diseases/medications which could influence the outcome of the therapy (e.g. uncontrolled diabetes mellitus, non-plaque-induced gingival diseases, antiepileptic drugs (phenytoin and sodium valproate), certain calcium channel-blocking drugs (e.g., nifedipine, verapamil, diltiazem, amlodipine, felodipine), immunoregulating drugs (e.g., ciclosporine), and high-dose oral contraceptives).
* Pregnant or nursing women.
* Presence of tooth mobility ≥ class 2.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-14 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Pocket closure | 5 years
  Defined as Probing pocket depth of 3 mm or less or Probing pocket depth of 4 mm with the absence of Bleeding on Probing in sites with Probing pocket depth of 6 mm or more at baseline.

SECONDARY OUTCOMES:
Tooth Retention | 5 years
  Number of teeth in the treated sextant will be calculated.
Number of instrumentation re-intervention | 5 years
  Number of instrumentation re-intervention during supportive periodontal therapy will be calculated
Mean Probing Pocket Depth changes | 5 years
  Defined as the mean changes in Probing pocket depth (distance in mm from the gingival margin to the bottom of the probable sulcus) at the involved sextant with respect to baseline.
Mean Clinical Attachment Level changes | 5 years
  Defined as the mean changes in Clinical Attachment Level (distance in mm from the Cemento Enamel Junction to the bottom of the probable sulcus) at the involved sextant with respect to baseline.
Mean recession changes | 5 years
  Defined as the changes in recession (distance in mm from Cemento Enamel Junction to the gingival margin).

OTHER OUTCOMES:
Discomfort during surgery | Immediately after surgery.
  Self reported on a 100-mm visual analog scale scale.